CLINICAL TRIAL: NCT03735498
Title: Psychological Intervention for Caregivers of Patients With Malignant Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Palliative Care Research Cooperative Group (Network)
Responsible Party: Principal Investigator, Deborah A Forst, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-426; U24NR014637 (NIH)
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Malignant Glioma
Keywords: Malignant Gliomas
MeSH Terms: conditions — Glioma | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological Intervention (Experimental): * Qualitative interview will be conducted
  * 7-item Generalized Anxiety Disorder measure will be completed by participants via mail correspondence or online
  * A psychoeducational component to address preparedness, manage expectations, and develop caregiving skills
  * A psychosocial component focusing on coping strategies, mindfulness, and facilitating acceptance while living with uncertainty
  * A self-care component to promote caregiver health and well-being
  Interventions: Other: Psychological Intervention

INTERVENTIONS:
Other: Psychological Intervention — Promote effective coping and reduce caregiving burden

SUMMARY:
This research study is evaluating a psychological intervention for caregivers of loved ones with malignant gliomas.

DETAILED DESCRIPTION:
Caregivers of loved ones with malignant gliomas frequently experience a physical and psychological burden caring for their loved ones. The purpose of this study is to find out whether a psychological intervention can help caregivers learn effective coping methods during their loved one's treatment and make the experience of being a caregiver more manageable.

The psychological intervention will take place in a series of six sessions. A trained social worker or psychologist will meet with the participant or talk with the participant over the telephone or by video conference for 45 minutes at a time to discuss the caregiver experience while developing effective skills to support the loved one as well as the participant over the course of the loved one's illness.

Upon the completion of the sessions, the investigators will have a short (30-minute) exit interview to obtain the participant's feedback on the intervention. The investigators will use the feedback to improve the intervention before further testing its effectiveness in future research studies. The investigators will also ask the participant to complete questionnaires before and after their participation in the intervention to help the investigators understand the participant's coping skills, caregiving burden, mood, and understanding about the loved one's illness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Identified by a patient with a malignant glioma (WHO Grade III or IV glioma) as the patient's primary caregiver
* The patient is receiving care at the MGH Cancer Center
* The patient was diagnosed with a malignant glioma within the past 6 months
* Able to speak and read in English
* Generalized Anxiety Disorder 7-item (GAD-7) score ≥5
* Participants may or may not be pregnant.

Exclusion Criteria:

* Deemed inappropriate for the study by the patient's clinician or the study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Forst, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mass General Hospital Cancer Center from February 2019 through October 2019. Interested participants were screened for eligibility using the GAD-7 tool with eligible participants having a score of 5 or greater.
Groups:
- Psychological Intervention: * 6 one-hour video conference sessions with mental health provider
  * participants complete survey battery before and after participating in the intervention
  * semi-structured interviews to assess acceptability of intervention
  Psychological Intervention: Promote effective coping and reduce caregiving burden
Period: Overall Study
Arm/Group | Psychological Intervention
Started | 13 (Total subjects who provided consent and were eligible to participate.)
Started Intervention | 10
Completed | 8 (Subjects who completed all 6 sessions.)
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Two participants did not complete all 6 sessions | 2

BASELINE CHARACTERISTICS:
Arm/Group | Psychological Intervention
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Caregiver Enrollment in the Intervention: Percentage of Eligible Caregivers Who Agree to Participate in the Study of This Intervention
Description: The investigators will report the percentage of eligible caregivers who agree to participate in the study of this intervention. The intervention will be deemed feasible if at least 70% (+/- 18%) of eligible caregivers are enrolled in the study.
Time Frame: 2 years
Population: We approached 30 potentially eligible caregivers of whom 21 provided consent to participate. Fourteen of those 21 patients met eligibility criteria based on the GAD-7 with one participant withdrawing consent prior to study enrollment. 13 of those 21 patients were able to proceed with the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Psychological Intervention
Number analyzed (Participants) | 30
Participants | 21

2. Primary Outcome: Feasibility of Caregiver Participation in a Population-specific Psychological Intervention: Percentage of Eligible Caregivers Who Participate in Each Session
Description: The investigators will report the percentage of eligible caregivers who participate in each session. Participation will be considered feasible if at least 70% of enrolled participants complete ≥50% of the sessions.
Time Frame: 2 years
Population: We evaluated the percentage of the 13 caregivers enrolled in the study that completed at least 50% of intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Psychological Intervention
Number analyzed (Participants) | 13
Participants | 10

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Psychological Intervention
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03735498/Prot_SAP_000.pdf